CLINICAL TRIAL: NCT05049564
Title: A Randomized Controlled Study of Microsurgical Clipping Via Keyhole Approaches Versus Traditional Open Approaches and Endovascular Coiling for Ruptured Anterior Circulation Aneurysms
Brief Title: Comparison of Clipping Via Keyhole Versus Traditional Approaches and Coiling for Ruptured Aneurysms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ZhuQing (Other)
Responsible Party: Sponsor-Investigator, ZhuQing, Chief Neurosurgeon, Second Affiliated Hospital of Soochow University
Organization: Second Affiliated Hospital of Soochow University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SJWKvascular001
Record Dates: First submitted 2021-08-31; First posted 2021-09-20 (Actual); Last update posted 2021-09-20 (Actual); Status verified 2021-09

CONDITIONS: Randomized Controlled Trial; Intracranial Aneurysm; Microsurgery; Endovascular Procedures
MeSH Terms: conditions — Intracranial Aneurysm

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- keyhole group (Experimental): patient harbored aneurysm who was treated by microsurgical clipping via keyhole approach.
  Interventions: Procedure: keyhole microneurosurgery
- conventional group (Experimental): patient harbored aneurysm who was treated by microsurgical clipping via conventional craniotomy.
  Interventions: Procedure: conventional microneurosurgery
- endovascular group (Experimental): patient harbored aneurysm who was treated by endovascular coiling via femoral approach.
  Interventions: Procedure: endovascular coiling

INTERVENTIONS:
Procedure: keyhole microneurosurgery — microsurgical clipping via keyhole approach
  Arms: keyhole group
Procedure: conventional microneurosurgery — microsurgical clipping via conventional craniotomy
  Arms: conventional group
Procedure: endovascular coiling — endovascular coiling via femoral approach
  Arms: endovascular group

SUMMARY:
Endovascular coiling has become a strategy of choice of intracranial aneurysms due to its minimally invasiveness. However, there has few prospective randomized controlled studies on the comparison of therapeutic effect between endovascular coiling and microsurgical clipping, especially the latter via keyhole approaches, which has been widely used in recent years. Based on the data of a single center, a randomized controlled study was conducted on patients with ruptured anterior circulation aneurysms suitable for both endovascular and extravascular treatment, including endovascular coiling, microsurgical clipping via conventional craniotomy and keyhole approaches, in order to compare the efficacy of the above strategies and provide more objective basis for treatment selection for operators.

DETAILED DESCRIPTION:
Consecutive patients of a single center will be screened. If spontaneous subarachnoid hemorrhage (SAH) is confirmed by head computed tomography (CT), a diagnostic CT angiography (CTA) or digital subtraction angiography (DSA) will be carried out emergently. A patients harbored a single intracranial aneurysm of anterior circulation that resulted in SAH will be concerned. Based on the assessment of condition, the patient will enrolled into this study without indication of decompressive craniectomy. The enrolled patients will be divided randomly into 3 groups, who experienced endovascular coiling, microsurgical clipping via conventional craniotomy and via keyhole approaches. All of these treatment will be conducted by a same senior neurosurgeon. CTA or DSA were followed up regularly. The occlusion rate, operative period, hospitalization duration and cost, surgical complications were compared and analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Single intracranial anterior circulation aneurysm diagnosed by CTA or DSA
* CT showed that subarachnoid hemorrhage originated from the rupture of the aneurysm and was confirmed during operation
* No indication of decompressive craniectomy (Hunt-Hess grade ≤ 4, Glasgow Coma Scale ≥ 7, no brain herniation; CT showed midline displacement < 5mm)
* The aneurysm is suitable for both endovascular treatment and microsurgical clipping

Exclusion Criteria:

* The patients and their families did not agree to join the study
* Patients with unruptured anterior circulation aneurysms
* Patients with posterior circulation aneurysms
* Patients with multiple intracranial aneurysms
* Those who cannot receive treatment due to serious concomitant diseases

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2013-01-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
occlusion rate of aneurysm | an average of 1 month
  occlusion rate of aneurysm
operative time | an average of 1 month
  total operative duration
hospitalization time | up to 3 months after discharge
  hospitalization duration
hospitalization cost | up to 3 months after discharge
  cost during hospitalization
postoperative complication rate | up to 3 months after discharge
  complication rate after intervention

SECONDARY OUTCOMES:
recurrent rate of aneurysm | 6 months after treatment
  recurrent rate after treatment of aneurysm
long-term complication rate | 6 months after treatment
  complication rate during follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Qing Lan, Doctor, Study Director — Second Affiliated Hospital of Soochow University

IPD SHARING:
Plan to Share IPD: No